CLINICAL TRIAL: NCT01098383
Title: Treatment With Acetyl-Choline Esterase Inhibitors in Children With Autism
Brief Title: Treatment With Acetyl-Choline Esterase Inhibitors in Children With Autism Spectrum Disorders
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sheba Medical Center (Other Government)
Collaborators: The Israeli Society of Clinical Pediatrics (HIPAK) (Unknown)
Responsible Party: Principal Investigator, Dr. Lidia Gabis MD, Dr. Lidia Gabis, Sheba Medical Center
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SHEBA-09-7151-LG-CTIL
Record Dates: First submitted 2010-03-11; First posted 2010-04-02 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Autism
Keywords: Autism
MeSH Terms: conditions — Autistic Disorder | interventions — Choline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo for AChEI and Choline (Placebo Comparator)
  Interventions: Drug: Indistinguishable placebo tablets, matching both donepezil and choline
- AChEI and Choline (Experimental): Acetyl-choline Esterase Inhibitor and Choline supplements
  Interventions: Drug: Acetyl-Choline Esterase Inhibitors and Choline supplements

INTERVENTIONS:
Drug: Acetyl-Choline Esterase Inhibitors and Choline supplements — Donepezil will be used at initial dose of 2.5 mg/day (during the first two weeks), and an increased dose of 5 mg/day (from the 3rd week and on), according to the treatment protocol listed below. The tablets will be taken during breakfast.
  AChE inhibitors are considered as potent agents for clinical use in Alzheimer's and Parkinson's dementias (Wevers & Schroder, 1999) and treatment with these agents was proven to be well-tolerated, safe and effective in these populations. Cholinergic side effects are generally transient, mild and dose-related, and primarily include diarrhea, nausea, and vomiting.
  Choline tablets will be taken at daily doses of 250 mg (in children with up to 40 kg body weight) and 500 mg (in children with more than 40 kg body weight), based on half of the adult daily dose.
  Arms: AChEI and Choline
Drug: Indistinguishable placebo tablets, matching both donepezil and choline — Indistinguishable placebo tablets, matching both donepezil and choline, will be given in the same amounts and schedules
  Arms: Placebo for AChEI and Choline

SUMMARY:
We propose a study which will combine multiple modalities in evaluating the treatment response of children with autism spectrum disorders (ASD) to acetyl-choline esterase (AChE) inhibitors and choline supplements. The primary objective of the study is to examine the efficacy of this treatment in improving core autistic symptoms. The Secondary objective of the study is to evaluate the safety and tolerability of the treatment protocol in ASD children. Exploratory objectives include evaluation of the influence of the treatment on linguistic performance, comorbid behaviors, adaptive functioning and executive functions.

DETAILED DESCRIPTION:
Autism Spectrum Disorders (ASD) are a group of developmental disorders of brain function resulting in a distinct phenotype, most probably related to many specific causes. Individuals with a disorder in the autism spectrum are a heterogeneous group of patients with early childhood onset of deficits in social interaction, communication and language, and repetitive and stereotypic behaviors. ASD has become increasingly prevalent during the last few decades (Wiznitzer, 2005).

The neuro-anatomical substrate of ASD has been the subject of intense investigation, but current findings are inconclusive, limited and sometimes even contradictory.

Medical treatment of autism is still a matter of dispute. Medications used are mainly aimed to treat the comorbid symptoms, such as epilepsy, tics, obsessive-compulsive or hyperactive behaviors (Wiznitzer, 2005). Although many efforts were invested in establishing a model of autistic pathophysiology, no such model is currently accepted, and there is no evidence for an efficient treatment of the core autistic symptoms (Wiznitzer, 2005).

Previous studies indicate that many brain systems are involved in the expression of autism. Specifically, it has been suggested that autism involves neurotransmitter dysregulations (Lam et al, 2006). A recent investigation of the cholinergic system in autism, detailed below, has provided promising findings. Our study aims to assess the clinical outcomes associated with cholinergic manipulations using pharmacological agents and nutritional supplements. The study approved by the Helsinki committee for clinical research.

ELIGIBILITY:
Inclusion criteria:

* A formal diagnosis of Autism or Pervasive Developmental Disorder not otherwise specified (PDD-NOS), given by a child neurologist.
* Age: 10-18 years.
* A signed parental consent form.

Exclusion criteria:

* Evidence for one of the following conditions:

  * an underlying infectious disease
  * chromosomal abnormality
  * metabolic disorder
  * specific brain related disorder (such as tuberous sclerosis)
  * history of fetal cytomegalovirus infection
  * birth asphyxia
  * a history of major head injury
  * a chronic use of non-steroidal anti-inflammatory drugs, (NSAID)
  * known brain damage
* Epilepsy
* Abnormal Electro-cardiogram (ECG)
* Epileptiform EEG
* Use of psychostimulants, anti-depressants, neuroleptics or anti-convulsive agents within the past month.
* Lack of cooperation in the screening phase

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 84 (Estimated)
Dates: Start 2010-03; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Core autistic symptoms (ATEC) | Once every 4 weeks during the first three mounth
  The parents will fill out this questionnaire about their child once every 4 weeks during the first Phase (12 weeks)- the Treatment phase.
Side effects and adverse events questionnaire | Once every 4 weeks during the first phase(12 weeks)
  A detailed parent questionnaire to assess side effects and adverse events. The parents will fill out these questionnaires about their child once every 4 weeks during the first phase(12 weeks)- which is the treatment phase.

SECONDARY OUTCOMES:
Linguistic performance (CELF-4) | After 6 mounth of washout
  The subject will be diagnosed on his Linguistic performance - using the CELF-4 diagnosis.
Adaptive functioning (Vineland-II) | After 6 mounth of washout
  The parents will be interviwed using the Adaptive functioning (Vineland-II)
Comorbid behaviors (CSI-4 questionnaire) | After 6 mouth of washout
  The parents will fill out the Comorbid behaviors (CSI-4) questionnaire
Executive functions (BRIEF questionnaire) | After 6 mounth of washout
  The parents will fill out the Executive functions (BRIEF) questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Lidia Gabis, MD, Principal Investigator — Sheba Medical Center; Dorit Ben-Shalom, Ph.D, Study Director — Ben-Gurion University of the Negev; Shefer Shahar, Dr., Study Director — Sheba Medical Center; Rotem Chayu Ben-Hur, MA, Study Director — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Ramat Gan, Israel

REFERENCES:
- [Derived] Iffland M, Livingstone N, Jorgensen M, Hazell P, Gillies D. Pharmacological intervention for irritability, aggression, and self-injury in autism spectrum disorder (ASD). Cochrane Database Syst Rev. 2023 Oct 9;10(10):CD011769. doi: 10.1002/14651858.CD011769.pub2. PMID 37811711
- [Derived] Ure A, Cox GR, Haslam R, Williams K. Acetylcholinesterase inhibitors for autistic spectrum disorders. Cochrane Database Syst Rev. 2023 Jun 1;6(6):CD013851. doi: 10.1002/14651858.CD013851.pub2. PMID 37267443